CLINICAL TRIAL: NCT06829511
Title: BARRIERS TOWARDS PHYSICAL ACTIVITY IN CARDIAC PATIENTS
Brief Title: BARRIERS TOWARDS PHYSICAL ACTIVITY
Acronym: CARDIAC PATIEN
Status: Not yet recruiting | Type: Observational
Sponsor: Bahria University (Other)
Responsible Party: Principal Investigator, Rabia Khan, Physiotherapist, Bahria University
Other Study IDs: BUHS-IRB # 114/24
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Cardiac Patients
MeSH Terms: interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire and Physical Exam — Cardiac Self-Efficacy Scale (CSES) 36-Item Short Form Survey (SF-36) Symptom Distress Scale (SDS)

SUMMARY:
A cross-sectional study of 323 cardiac patients aged 40 to 60 will be carried out at PNS Shifa and the National Institute of Cardiovascular Diseases. Data will be gathered using surveys and evaluated with SPSS software. The results are likely to show considerable differences in barrier frequency across demographic groups, offering insights into targeted treatments.

Understanding these limitations is critical for establishing successful physical activity regimens, improving heart health, and, eventually, lowering rehospitalization rates. The findings will help to develop specific approaches to overcome these challenges and encourage regular physical exercise among cardiac patients.

Objectives:

1. To identify and categorize the specific barriers to physical activity faced by cardiac patients.
2. To analyze how these barriers differ among various demographic groups (e.g., age, gender).
3. To examine how barriers to physical activity vary according to clinical characteristics.

Methodology:

Using a cross sectional study design, data data was collected from NICVD hospital and PNS shifa hospital by providing questionnaires to patient having cardiac disease. The questionnaires comprises of close ended questions.

ELIGIBILITY:
Inclusion Criteria:

* 1. Heart patients who have been diagnosed with a cardiovascular condition for more than six months.

  2. People between the ages of forty and sixty. 3. It was acceptable to have both male and female participants. 4. Patients either already participating in a cardiac rehabilitation program or those who had yet to engage in one were included.

Exclusion Criteria:

1. Existence of musculoskeletal disorders that might affect their physical activity levels.
2. Neurological conditions that could hinder exercise participation or influence responses to surveys.
3. Chronic illnesses such as diabetes or irritable bowel syndrome that could interfere with the barriers evaluated in the study.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: cardiac patients
Sampling Method: Non-Probability Sample
Enrollment: 323 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
risk factors | 2 weeks
  We will recurit cardiac patients with the questioonare for the risk factors and reasons not to engage in physical activity

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sutherland S, Penfold R, Doherty A, Milne Z, Dawes H, Pugh C, Boulton M, Newton JL. A cross-sectional study exploring levels of physical activity and motivators and barriers towards physical activity in haemodialysis patients to inform intervention development. Disabil Rehabil. 2021 Jun;43(12):1675-1681. doi: 10.1080/09638288.2019.1672214. Epub 2019 Oct 24. PMID 31646910